CLINICAL TRIAL: NCT05790200
Title: A Phase II Clinical Study of Cadonilimab (AK104) Combined With Chemotherapy in the Treatment of PD-1 Inhibitor Resistant Nasopharyngeal Carcinoma
Brief Title: Cadonilimab (AK104) in the Treatment of Nasopharyngeal Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, kunyu yang, Chief physician, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: AK104-IIT
Record Dates: First submitted 2023-03-01; First posted 2023-03-30 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cadonilimab (AK104) combined with chemotherapy (Experimental): Cadonilimab (200 mg, administered on the first day of each cycle, Q3W, until there is no clinical benefit)+platinum-based chemotherapy, Q3W, 4-6 cycles), every 3 weeks (21 days) is a treatment cycle
  Interventions: Drug: Cadonilimab

INTERVENTIONS:
Drug: Cadonilimab — Cadonilimab (200 mg, administered on the first day of each cycle, Q3W, until there is no clinical benefit)+platinum-based chemotherapy, Q3W, 4-6 cycles), every 3 weeks (21 days) is a treatment cycle.
  Other Names: AK104

SUMMARY:
This study is a phase II clinical study of Cadonilimab (AK104) combined with chemotherapy in the treatment of PD-1 inhibitor-resistant nasopharyngeal carcinoma.

DETAILED DESCRIPTION:
The purpose is to evaluate the safety and effectiveness of Cadonilimab combined with chemotherapy in the treatment of PD-1 inhibitor-resistant nasopharyngeal carcinoma as the second line and above. This study is a single-arm, phase II clinical study. It is planned to enroll about 30 patients with PD-1 inhibitor resistant nasopharyngeal carcinoma. PD-Ll CPS (<50% vs>50%, subjects whose PD-Ll expression could not be evaluated were classified as<50%) was used as the stratification factor. The study will set up a safety induction period. It is planned to enroll about 6 PD-1 inhibitor resistant subjects first, and the researchers will conduct a preliminary safety assessment. If the safety and tolerability are good, and the preliminary curative effect signal is observed, it will enter the extended group period. When about 15 subjects are selected, effectiveness analysis will be carried out. If 6 of the 15 subjects with severe side effects can not tolerate, the researcher may stop the group of subjects after discussion. In case of poor safety, the researcher decided to revise or stop the study after discussion.

ELIGIBILITY:
Inclusion Criteria:

1. The age at the time of enrollment is more than 18 years old and less than 75 years old, both male and female.
2. The Eastern Cancer Cooperation Organization (ECOG) physical fitness score was 0 or 1.
3. The expected survival period is more than 3 months.
4. Nasopharyngeal carcinoma confirmed by histology or cytology.
5. The subject has previously received treatment with PD-1 inhibitor and failed without indication of radical local treatment.

According to the evaluation standard of curative effect of solid tumor, RECIST v l L At least one measurable lesion.

Exclusion Criteria:

1. Except for nasopharyngeal carcinoma, the subjects had other malignant tumors within 2 years before enrollment. Subjects with other tumors that have been cured by local treatment, such as basal or cutaneous squamous cell carcinoma, superficial bladder cancer, cervical or breast cancer in situ, are not excluded.
2. He participated in the treatment of experimental drugs within 4 weeks before the first study administration.
3. Patients with active autoimmune diseases that require systematic treatment in the past two years (such as the use of disease improvement drugs, corticosteroids, immunosuppressive therapy), and replacement therapy (such as thyroxine, insulin, or physiological corticosteroid replacement therapy for adrenal or pituitary insufficiency) are not considered as a systemic treatment.
4. Have a history of immune deficiency; HIV antibody test positive; At present, systemic corticosteroids or other immunosuppressants are being used for a long time.
5. Active tuberculosis (TB) is known. Subjects suspected of active TB should be excluded from active TB.
6. The history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation are known.
7. The untreated active hepatitis B subjects (HBsAg positive and HBV-DNA more than 1000 copies/ml (200 IU/ml) or higher than the lower detection limit, whichever is higher) are required to receive anti hepatitis B virus treatment during the study treatment period; Active hepatitis C subjects (HCV antibody positive and HCV-RNA level higher than the lower limit of detection).
8. Major surgical operation or serious injury occurred within 30 days before the first administration, or major surgical operation planner (determined by the researcher) within 30 days after the first administration; Minor local operations (excluding central venous catheterization via peripheral vein puncture) were performed within 3 days before the first administration.
9. There is central nervous system metastasis.
10. There are currently uncontrolled concomitant diseases, including but not limited to symptomatic congestive heart failure (grade 2 and above determined according to the functional classification of the New York Heart Association), unstable angina pectoris, acute myocardial ischemia, poorly controlled arrhythmia, decompensated liver cirrhosis, nephrotic syndrome, uncontrolled metabolic disorder, severe active peptic ulcer disease or gastritis, Mental illness/social condition that may limit the subject's compliance with the research requirements or affect the subject's ability to provide written informed consent.
11. There was a history of myocarditis, cardiomyopathy and malignant arrhythmia in the past. Unstable angina pectoris, congestive heart failure or vascular disease (such as aortic aneurysm or peripheral venous thrombosis requiring surgical repair) that needs hospitalization within 12 months before the first administration of the drug, or other cardiac damage that may affect the safety evaluation of the study drug (such as poorly controlled arrhythmia, myocardial infarction or ischemia); There is a history of esophageal and gastric varices, serious ulcer, wound healing, gastrointestinal perforation, abdominal pain, gastrointestinal obstruction, abdominal abscess or acute gastrointestinal bleeding within 6 months before the first administration; Any arterial thromboembolic event occurred within 6 months before the first administration, including venous thromboembolic generation of NC I CTCAE 5.0 grade 3 and above, transient ischemic attack, cerebrovascular accident, hypertensive crisis or hypertensive encephalopathy; Acute exacerbation of chronic obstructive pulmonary disease occurred within 1 month before the first administration; There is currently hypertension and after treatment with oral antihypertensive drugs, the systolic blood pressure is more than 160 mmHg or the diastolic blood pressure is less than 100 mmHg.
12. Have a history of severe bleeding tendency or coagulation dysfunction; One month before the first administration, there were blood symptoms with significant clinical significance, including but not limited to gastrointestinal bleeding, hemoptysis, screening imaging showed that the tumor wrapped around important blood vessels or had obvious necrosis and cavity, and the researcher believed that participating in the study might cause bleeding risk;
13. The toxicity of previous anti-tumor treatment has not been relieved, which is defined as that the toxicity has not returned to the level 0 or 1 of NC l CTCAE 5.0, or the level specified in the inclusion/exclusion criteria, except for the sequelae of hair loss and previous lead treatment related neurotoxicity. Subjects (such as hearing loss) who have irreversible toxicity and are not expected to worsen after administration of the study drug may be included in the study after consultation with the medical examiner. Subjects with long-term toxicity caused by radiotherapy that cannot be recovered according to the judgment of the researcher may be included in the study after consultation with the medical supervisor.
14. The live vaccine was vaccinated within 30 days before the first administration, or was planned to be vaccinated during the study period.
15. Known allergy to any component of any study drug; A history of severe hypersensitivity to other monoclonal antibodies is known.
16. Known history of mental illness, drug abuse, alcohol or drug abuse.
17. Pregnant or lactating women.
18. Any previous or current disease, treatment, or laboratory test abnormality may confuse the results of the study, affect the full participation of the subject in the study, or participation in the study may not be in the best interests of the subject.
19. Local or systemic diseases caused by non-malignant tumors, or diseases or symptoms secondary to tumors, which can lead to higher medical risk and/or uncertainty of survival evaluation, such as tumor-like leukemia reaction (white blood cell count>20 X 109/L or cachexia performance (such as known weight loss of more than 10% in the 3 months before screening), etc

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2025-09-22 (Estimated); Study Completion 2025-09-22 (Estimated)

PRIMARY OUTCOMES:
Adverse Event(AE) | From randomization to the end of the study，the evaluation lasts for 24 months
  The type, frequency, severity, timing, seriousness, and relationship to study therapyclinical significance
Objective Response Rate，ORR | The last subject completes at least 24 weeks of follow-up (or disease progression)
  The proportion of patients whose tumor volume is reduced to 30% and can be maintained for more than 4 weeks,Based on RECIST v i I Assessed ORR
Progression-free survival，PFS | The last subject completes at least 24 weeks of follow-up (or disease progression)
  The time from the beginning of the patient's treatment to the disease progression or death for any reason.Based on RECIST v i I Assessed PFS

SECONDARY OUTCOMES:
Overall Survival,OS | 3 years
  The time from the patient receiving treatment to the death of the patient for any reason,OS evaluated according to RECIST vi. I

OTHER OUTCOMES:
Time to progress，TTP | The last subject completes at least 24 weeks of follow-up (or disease progression)
  The time from the beginning of the patient's treatment to the occurrence and progression of the tumor

CONTACTS AND LOCATIONS:
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2022-09-18): https://cdn.clinicaltrials.gov/large-docs/00/NCT05790200/Prot_000.pdf